CLINICAL TRIAL: NCT04088565
Title: Mechanisms of Non-invasive Vagus Nerve Stimulation Underlying Enhanced Motor Control in Humans
Brief Title: VNS-induced Corticospinal Plasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, George Wittenberg, Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY19040394 (Aim 1)
Record Dates: First submitted 2019-09-09; First posted 2019-09-13 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Stroke
Keywords: Neuromodulation; Paresis; Neurorehabilitation
MeSH Terms: conditions — Stroke; Paresis | interventions — Vagus Nerve Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PAS+VNS (Experimental): Paired-associative stimulation (PAS) targeting primary motor cortex will be administered with VNS in individuals with hemiparesis secondary to stroke and neurologically-intact, age-matched controls.
  Interventions: Other: Paired-Associative Stimulation (PAS); Other: Vagus Nerve Stimulation (VNS)
- PAS+Sham (Sham Comparator): Paired-associative stimulation (PAS) targeting primary motor cortex will be administered with sham stimulation in individuals with hemiparesis secondary to stroke and neurologically-intact, age-matched controls.
  Interventions: Other: Paired-Associative Stimulation (PAS); Other: Sham Stimulation

INTERVENTIONS:
Other: Paired-Associative Stimulation (PAS) — Simultaneous activation of connections in motor cortex via stimulation to the nerves and brain.
  Other Names: PAS
Other: Vagus Nerve Stimulation (VNS) — Recruits the auricular branch of the vagus nerve which activates brain structures that release chemicals mediating cortical plasticity.
  Other Names: VNS
  Arms: PAS+VNS
Other: Sham Stimulation — Sub-threshold stimulation that does not activate neural structures.
  Other Names: Sham
  Arms: PAS+Sham

SUMMARY:
The goal of this study is to learn more about the connections between the brain, spinal cord, and muscles and how these connections can be strengthened after neurological injury.

DETAILED DESCRIPTION:
Non-invasive stimulation techniques can be used to appropriately time converging inputs to induce changes in cortical output circuits of human primary motor cortex, a neuromodulatory protocol known as paired-associative stimulation (PAS). Experiments seek to examine interactions between cortical PAS and non-invasive vagus nerve stimulation (VNS) to understand the extent to which VNS amplifies cortical plasticity in humans.

ELIGIBILITY:
Inclusion Criteria:

INDIVIDUALS WHO HAVE HAD A STROKE:

1. Diagnosis of first ever stroke
2. At least 6 months after stroke onset
3. Motor-evoked potentials in hand/arm muscles
4. Subjects must show an understanding of the study goals and have the ability to follow simple directions as judged by the investigators.

   ALL INDIVIDUALS:
5. Between the ages of 18 and 75 years old

Exclusion Criteria:

INDIVIDUALS WHO HAVE HAD A STROKE:

1. Hemispatial neglect, aphasia, or cognitive impairment that would impact testing and would interfere with the ability to follow simple instructions, as judged by the investigators

   ALL INDIVIDUALS:
2. Neurological disorder(s) influencing movement (besides stroke)
3. History of seizure or epilepsy
4. Metallic brain implants
5. Bodily implants such as cardioverter defibrillators, insulin pumps, ventriculoperitoneal shunts, cochlear implants, or pacemakers
6. Pregnant or expecting to become pregnant
7. Difficulty maintaining alertness and/or remaining still
8. Silicone or plastic allergy
9. History of vestibular disorders (eg, Vertigo, Meniere's Disease, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2021-11-09 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Change in size of evoked potential | 1 week
  The primary endpoint is the change from baseline (ie, before PAS) in the size of evoked potentials. Differences in the change between conditions (ie, PAS+VNS vs PAS+Sham) will address whether VNS drives cortical plasticity.

CONTACTS AND LOCATIONS:
Overall Officials: George F Wittenberg, MD, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team may share data with scientists at other centers for the purpose of data analysis and collaboration. Research information and data may be shared with investigators conducting other research. This information will not be identifiable.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Information may be shared while data is being recorded, analyzed, and/or prior to publication. Data may be available for seven years after manuscripts are published.
Access Criteria: Data use agreements will be established with scientists at other centers, or conducting other research, prior to any data sharing.

REFERENCES:
- [Background] Nakayama H, Jorgensen HS, Raaschou HO, Olsen TS. Recovery of upper extremity function in stroke patients: the Copenhagen Stroke Study. Arch Phys Med Rehabil. 1994 Apr;75(4):394-8. doi: 10.1016/0003-9993(94)90161-9. PMID 8172497
- [Background] Pollock A, St George B, Fenton M, Firkins L. Top ten research priorities relating to life after stroke. Lancet Neurol. 2012 Mar;11(3):209. doi: 10.1016/S1474-4422(12)70029-7. No abstract available. PMID 22341029
- [Background] Langhorne P, Coupar F, Pollock A. Motor recovery after stroke: a systematic review. Lancet Neurol. 2009 Aug;8(8):741-54. doi: 10.1016/S1474-4422(09)70150-4. PMID 19608100
- [Background] Heidenreich PA, Trogdon JG, Khavjou OA, Butler J, Dracup K, Ezekowitz MD, Finkelstein EA, Hong Y, Johnston SC, Khera A, Lloyd-Jones DM, Nelson SA, Nichol G, Orenstein D, Wilson PW, Woo YJ; American Heart Association Advocacy Coordinating Committee; Stroke Council; Council on Cardiovascular Radiology and Intervention; Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Arteriosclerosis; Thrombosis and Vascular Biology; Council on Cardiopulmonary; Critical Care; Perioperative and Resuscitation; Council on Cardiovascular Nursing; Council on the Kidney in Cardiovascular Disease; Council on Cardiovascular Surgery and Anesthesia, and Interdisciplinary Council on Quality of Care and Outcomes Research. Forecasting the future of cardiovascular disease in the United States: a policy statement from the American Heart Association. Circulation. 2011 Mar 1;123(8):933-44. doi: 10.1161/CIR.0b013e31820a55f5. Epub 2011 Jan 24. PMID 21262990
- [Background] Porter BA, Khodaparast N, Fayyaz T, Cheung RJ, Ahmed SS, Vrana WA, Rennaker RL 2nd, Kilgard MP. Repeatedly pairing vagus nerve stimulation with a movement reorganizes primary motor cortex. Cereb Cortex. 2012 Oct;22(10):2365-74. doi: 10.1093/cercor/bhr316. Epub 2011 Nov 10. PMID 22079923
- [Background] Khodaparast N, Hays SA, Sloan AM, Hulsey DR, Ruiz A, Pantoja M, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation during rehabilitative training improves forelimb strength following ischemic stroke. Neurobiol Dis. 2013 Dec;60:80-8. doi: 10.1016/j.nbd.2013.08.002. Epub 2013 Aug 15. PMID 23954448
- [Background] Khodaparast N, Hays SA, Sloan AM, Fayyaz T, Hulsey DR, Rennaker RL 2nd, Kilgard MP. Vagus nerve stimulation delivered during motor rehabilitation improves recovery in a rat model of stroke. Neurorehabil Neural Repair. 2014 Sep;28(7):698-706. doi: 10.1177/1545968314521006. Epub 2014 Feb 18. PMID 24553102
- [Background] Meyers EC, Solorzano BR, James J, Ganzer PD, Lai ES, Rennaker RL 2nd, Kilgard MP, Hays SA. Vagus Nerve Stimulation Enhances Stable Plasticity and Generalization of Stroke Recovery. Stroke. 2018 Mar;49(3):710-717. doi: 10.1161/STROKEAHA.117.019202. Epub 2018 Jan 25. PMID 29371435
- [Background] Dawson J, Pierce D, Dixit A, Kimberley TJ, Robertson M, Tarver B, Hilmi O, McLean J, Forbes K, Kilgard MP, Rennaker RL, Cramer SC, Walters M, Engineer N. Safety, Feasibility, and Efficacy of Vagus Nerve Stimulation Paired With Upper-Limb Rehabilitation After Ischemic Stroke. Stroke. 2016 Jan;47(1):143-50. doi: 10.1161/STROKEAHA.115.010477. Epub 2015 Dec 8. PMID 26645257
- [Background] Kilgard MP, Rennaker RL, Alexander J, Dawson J. Vagus nerve stimulation paired with tactile training improved sensory function in a chronic stroke patient. NeuroRehabilitation. 2018;42(2):159-165. doi: 10.3233/NRE-172273. PMID 29562561
- [Background] Kimberley TJ, Pierce D, Prudente CN, Francisco GE, Yozbatiran N, Smith P, Tarver B, Engineer ND, Alexander Dickie D, Kline DK, Wigginton JG, Cramer SC, Dawson J. Vagus Nerve Stimulation Paired With Upper Limb Rehabilitation After Chronic Stroke. Stroke. 2018 Nov;49(11):2789-2792. doi: 10.1161/STROKEAHA.118.022279. PMID 30355189